CLINICAL TRIAL: NCT00247416
Title: Randomized Phase II Trail of Carboplatin and Gemcitabine Untreated Stage IIIB-pleural Effusion and Stage IV Lung Cancer
Brief Title: Effects of Carboplatin and Gemcitabine on Stage IIIB Pleural Effusion and Stage IV Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Susanne Arnold (Other)
Collaborators: Kentucky Lung Cancer Research Program (Other)
Responsible Party: Sponsor-Investigator, Susanne Arnold, Sponsor/Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTN-0501
Record Dates: First submitted 2005-10-28; First posted 2005-11-01 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-01

CONDITIONS: Stage IV Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer
Keywords: Untreated; Lung; Cancer; non-small cell; gemcitabine; gemzar; carboplatin; dexamethasone
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Gemcitabine; Dexamethasone; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 No Dex (Other): No Dexamethasone
  Interventions: Drug: Gemcitabine; Drug: Carboplatin
- 2 Dex (Experimental): Dexamethasone
  Interventions: Drug: Gemcitabine; Drug: Dexamethasone; Drug: Carboplatin

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 intravenously over 30 minutes on days 5 and 12.
  Other Names: Gemzar
Drug: Dexamethasone — 16 mg bid for 4 days prior to each chemotherapy start.
  Arms: 2 Dex
Drug: Carboplatin — AUC 6.0 intravenously over 30 minutes on day 5.

SUMMARY:
The purpose of this study is to find better treatment for lung cancer and to find out what effects the combined treatment of carboplatin and gemcitabine when given with or without dexamethasone have on cancer.

This study will determine if dexamethasone, when given before standard chemotherapy will increase the cancer fighting effects and reduce the side effects of chemotherapy.

DETAILED DESCRIPTION:
Subjects enrolled in the study will be placed in one of two treatment arms. All subjects have a 50-50 chance of being placed into either treatment arm. Treatment Arm 1 will receive chemotherapy alone, Treatment Arm 2 will receive chemotherapy with dexamethasone given pre-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Untreated, stage IIIB with pleural effusion
* Untreated, Stage IV, non-small cell lung cancer
* Recurrent after surgery if no previous radiation therapy or chemotherapy were administered as part of their primary treatment, except for palliative radiotherapy
* 18 years of age or older
* ECOG PS 0, 1 or 2
* At Least one target lesion according to the RECIST Criteria
* Adequate organ and marrow function

Exclusion Criteria:

* Previous cancer history unless they have had curative treatment completed at least 5 years prior to entry.
* No previous radiotherapy, chemotherapy or immunotherapy for NSCLC, except for radiation therapy to the brain to control metastasis, bone to control pain, or lung to relieve bronchial obstruction.
* No radiation therapy for any previous cancer to more than 25% of bone marrow.
* Uncontrolled, intercurrent illness
* Non-study corticosteroids
* Pregnant women
* Peripheral neuropathy greater than grade 1
* Uncontrolled seizures, central nervous system disorders
* Major surgery within 4 weeks of the start of study treatment
* Lack of complete recovery from major surgery.
* Glaucoma
* Lack of physical integrity of upper gastrointestinal tract, inability to swallow tablets
* Severe acquired or hereditary immunodeficiency
* Patients with brain metastases must receive definitive treatment (radiation, surgery or both) and be clinically and radiologically stable for 4 weeks & off corticosteroids for at least 2 weeks prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Rinehart, Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky
Locations (7):
- United States (7):
  - Commonwealth Cancer Center, Danville, Kentucky
  - Markey Cancer Center, Lexington, Kentucky
  - Brown Cancer Center, Louisville, Kentucky
  - St. Claire Regional Medical Center, Morehead, Kentucky
  - Montgomery Cancer Center, Mount Sterling, Kentucky
  - Owensboro Medical HealthCare System, Owensboro, Kentucky
  - West Kentucky Hematology & Oncology Group, PSC, Paducah, Kentucky

REFERENCES:
- [Result] Rinehart J, Arnold S, Kloecker G, Lim A, Zaydan MA, Baeker T, Maheshwari JG, Carloss H, Slone S, Shelton B, Croley J, Kvale E, Brooks M, Leggas M. Phase II randomized trial of carboplatin and gemcitabine with or without dexamethasone pre-treatment in patients with Stage IV non-small cell lung cancer. Cancer Chemother Pharmacol. 2013 May;71(5):1375-83. doi: 10.1007/s00280-013-2111-3. Epub 2013 Mar 9. PMID 23475103

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total number of patients enrolled is 60. However, 1 patient enrolled to trial was discontinued from trial prior to receipt of any study therapies; patient was randomized to arm 1 (control, no dexamethasone pretreatment) but received no study therapies or procedures.
Groups:
- Arm 1, Control, no Dexamethasone Pretreatment: Patients with stage 4 untreated non-small cell lung cancer received carboplatin (AUC 6, day 1) and gemcitabine (1000 mg/m2 days 1, 8) for up to 6 cycles with no dexamethasone pretreatment.
- Arm 2, Dexamethasone Pretreatment Test Arm: Patients with stage 4 untreated non-small cell lung cancer received carboplatin (AUC 6, day 1) and gemcitabine (1000 mg/m2 days 1, 8) for up to 6 cycles with dexamethasone pretreatment.Dexamethasone pretreatment = dexamethasone 16 mg, bid 4 days before and day of each chemotherapy treatment (days 1 and 8).
Period: Overall Study
Arm/Group | Arm 1, Control, no Dexamethasone Pretreatment | Arm 2, Dexamethasone Pretreatment Test Arm
Started | 26 | 33
Completed | 25 | 31
Not Completed | 1 | 2
Not completed — 3 patients were found to be ineligible | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1, Control, no Dexamethasone Pretreatment | Arm 2, Dexamethasone Pretreatment Test Arm | Total
Number analyzed (Participants) | 25 | 31 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 27 | 45
  >=65 years | 7 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 12 | 17 | 29
Region of Enrollment [Number; unit: participants]
  United States | 25 | 31 | 56

OUTCOME MEASURES:

1. Secondary Outcome: Effect of Dexamethasone Pre-treatment on Response Rate.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Pre-treatment, pre-cycles 3 & 5, and up to 4 weeks after last treatment
Measure: Number (95% Confidence Interval); unit: percentage of responders out of total
Arm/Group | 1 No Dex | 2 Dex
Number analyzed (Participants) | 25 | 31
percentage of responders out of total | 8 [0.1 to 26.0] | 26 [11.9 to 44.6]

2. Primary Outcome: Percentage of Participants With Reduction in Grade 3/4 Neutropenia
Description: Reduction grade 3/4 neutropenia
Time Frame: continuous throughout treatment, up to 25 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1, Control, no Dexamethasone Pretreatment | Arm 2, Dexamethasone Pretreatment Test Arm
Number analyzed (Participants) | 25 | 31
percentage of participants | 40 | 13

3. Secondary Outcome: Effect of Dexamethasone Pre-treatment on Overall Survival.
Description: Overall survival
Time Frame: Pre-treatment, pre-cycles 3 & 5,4 weeks after last treatment, every 3 months, an average of 471 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm 1, Control, no Dexamethasone Pretreatment | Arm 2, Dexamethasone Pretreatment Test Arm
Number analyzed (Participants) | 25 | 31
days | 291 [228 to 437] | 378 [189 to 608]

4. Secondary Outcome: Progression-free Survival
Description: progression-free survival
Time Frame: Pre-treatment, pre-cycles 3 & 5,4 weeks after last treatment, and every 3 months, an average of 471 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm 1, Control, no Dexamethasone Pretreatment | Arm 2, Dexamethasone Pretreatment Test Arm
Number analyzed (Participants) | 25 | 31
days | 101 [60 to 172] | 122 [82 to 185]

ADVERSE EVENTS:
Groups:
- 1 No Dexamethasone: Patients with stage 4 untreated non-small cell lung cancer received carboplatin (AUC 6, day 1) and gemcitabine (1000 mg/m2 days 1, 8) for up to 6 cycles with no dexamethasone pretreatment.
- 2 Dexamethasone: Patients with stage 4 untreated non-small cell lung cancer received carboplatin (AUC 6, day 1) and gemcitabine (1000 mg/m2 days 1, 8) for up to 6 cycles with dexamethasone pretreatment.Dexamethasone pretreatment = dexamethasone 16 mg, bid 4 days before and day of each chemotherapy treatment (days 1 and 8).
Arm/Group | 1 No Dexamethasone | 2 Dexamethasone
Serious Adverse Events (participants affected / at risk) | 7/26 | 12/33
Other Adverse Events (participants affected / at risk) | 26/26 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1 No Dexamethasone (N=26) | 2 Dexamethasone (N=33)
ANEMIA (Blood and lymphatic system disorders) | 0 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 2
HEART ARREST (Cardiac disorders) | 1 | 1
CONSTIPATION (Gastrointestinal disorders) | 2 | 0
DIARRHEA (Gastrointestinal disorders) | 0 | 1
DUODENAL ULCER (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 1
RECTAL DISORDER (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 0
MEDICATION ERROR (General disorders) | 0 | 1
SEPSIS (General disorders) | 0 | 3
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 0 | 1
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 1 | 0
URINARY TRACT INFECTION (Renal and urinary disorders) | 0 | 1
APNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
COUGH INCREASED (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 2 | 3
PULMONARY EMBOLUS (Respiratory, thoracic and mediastinal disorders) | 0 | 3
DEEP THROMBOPHLEBITIS (Vascular disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 0 | 1
MESENTERIC VENOUS OCCLUSION (Vascular disorders) | 0 | 1
THROMBOSIS (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1 No Dexamethasone (N=26) | 2 Dexamethasone (N=33)
ANEMIA (Blood and lymphatic system disorders) | 18 | 24
ECCHYMOSIS (Blood and lymphatic system disorders) | 3 | 0
HYPOCHROMIC ANEMIA (Blood and lymphatic system disorders) | 0 | 3
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 10
LEUKOPENIA (Blood and lymphatic system disorders) | 18 | 19
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 | 0
PETECHIA (Blood and lymphatic system disorders) | 3 | 0
THROMBOCYTHEMIA (Blood and lymphatic system disorders) | 0 | 5
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 18 | 24
TACHYCARDIA (Cardiac disorders) | 3 | 0
CUSHINGS SYNDROME (Endocrine disorders) | 0 | 3
CONJUNCTIVITIS (Eye disorders) | 0 | 2
ANOREXIA (Gastrointestinal disorders) | 5 | 9
CHOLECYSTITIS (Gastrointestinal disorders) | 2 | 0
CONSTIPATION (Gastrointestinal disorders) | 12 | 18
DIARRHEA (Gastrointestinal disorders) | 5 | 8
DYSPEPSIA (Gastrointestinal disorders) | 0 | 2
DYSPHAGIA (Gastrointestinal disorders) | 0 | 2
FLATULENCE (Gastrointestinal disorders) | 0 | 2
MOUTH ULCERATION (Gastrointestinal disorders) | 0 | 4
NAUSEA (Gastrointestinal disorders) | 16 | 20
ORAL MONILIASIS (Gastrointestinal disorders) | 0 | 5
RECTAL DISORDER (Gastrointestinal disorders) | 0 | 2
STOMATITIS (Gastrointestinal disorders) | 3 | 9
ULCERATIVE STOMATITIS (Gastrointestinal disorders) | 0 | 2
VOMITING (Gastrointestinal disorders) | 12 | 7
ABDOMINAL PAIN (General disorders) | 0 | 3
ACCIDENTAL INJURY (General disorders) | 2 | 0
ASTHENIA (General disorders) | 17 | 23
BACK PAIN (General disorders) | 2 | 3
CHEST PAIN (General disorders) | 3 | 6
FACE EDEMA (General disorders) | 0 | 2
FEVER (General disorders) | 7 | 5
HEADACHE (General disorders) | 2 | 3
INJECTION SITE PAIN (General disorders) | 3 | 0
INJECTION SITE REACTION (General disorders) | 2 | 0
LAB TEST ABNORMAL (General disorders) | 4 | 7
MUCOUS MEMBRANE DISORDER (General disorders) | 2 | 2
PAIN (General disorders) | 11 | 7
INFECTION FUNGAL (Infections and infestations) | 2 | 0
ALKALINE PHOSPHATASE INCREASED (Metabolism and nutrition disorders) | 0 | 2
BUN INCREASED (Metabolism and nutrition disorders) | 0 | 3
CREATININE INCREASED (Metabolism and nutrition disorders) | 0 | 3
DEHYDRATION (Metabolism and nutrition disorders) | 6 | 0
EDEMA (Metabolism and nutrition disorders) | 2 | 6
GOUT (Metabolism and nutrition disorders) | 2 | 0
HYPERCALCEMIA (Metabolism and nutrition disorders) | 0 | 3
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 4 | 14
HYPOCALCEMIA (Metabolism and nutrition disorders) | 0 | 3
HYPOKALEMIA (Metabolism and nutrition disorders) | 6 | 13
HYPONATREMIA (Metabolism and nutrition disorders) | 3 | 6
HYPOPROTEINEMIA (Metabolism and nutrition disorders) | 3 | 15
PERIPHERAL EDEMA (Metabolism and nutrition disorders) | 4 | 10
RESPIRATORY ALKALOSIS (Metabolism and nutrition disorders) | 0 | 2
SGOT INCREASED (Metabolism and nutrition disorders) | 2 | 7
SGPT INCREASED (Metabolism and nutrition disorders) | 2 | 8
WEIGHT LOSS (Metabolism and nutrition disorders) | 2 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 2
MYASTHENIA (Musculoskeletal and connective tissue disorders) | 0 | 5
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 2 | 0
ANXIETY (Nervous system disorders) | 2 | 3
CONFUSION (Nervous system disorders) | 0 | 2
DEPRESSION (Nervous system disorders) | 2 | 2
DIZZINESS (Nervous system disorders) | 2 | 4
HYPERTENSION (Nervous system disorders) | 3 | 2
INSOMNIA (Nervous system disorders) | 10 | 15
NEUROPATHY (Nervous system disorders) | 4 | 4
PARESTHESIA (Nervous system disorders) | 0 | 2
URINARY RETENTION (Nervous system disorders) | 0 | 2
VASODILATATION (Nervous system disorders) | 4 | 7
KIDNEY FUNCTION ABNORMAL (Renal and urinary disorders) | 0 | 2
URINARY TRACT INFECTION (Renal and urinary disorders) | 2 | 2
COUGH INCREASED (Respiratory, thoracic and mediastinal disorders) | 10 | 10
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 13 | 13
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 | 2
HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 4 | 0
HICCUP (Respiratory, thoracic and mediastinal disorders) | 0 | 2
HYPOVENTILATION (Respiratory, thoracic and mediastinal disorders) | 0 | 2
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 5 | 2
LUNG EDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 2
PHARYNGITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 4
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 2 | 4
RHINITIS (Respiratory, thoracic and mediastinal disorders) | 3 | 3
SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 5
RASH (Skin and subcutaneous tissue disorders) | 8 | 6
SWEATING (Skin and subcutaneous tissue disorders) | 0 | 7
HYPOTENSION (Vascular disorders) | 0 | 2
PALLOR (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No